CLINICAL TRIAL: NCT04141657
Title: Observational Prospective Multidirectional Study on the Safety of Antimicrobial Pharmacotherapy in Intensive Care Unit (ICU) Children Aged 0-17
Brief Title: Safety Analysis of Antimicrobial Pharmacotherapy in Intensive Care Unit at Pediatric Hospital
Status: Completed | Type: Observational
Sponsor: Anna Vlasova (Other Government)
Collaborators: Russian Medical Academy of Continuous Professional Education (Unknown); Morozov Children's Municipal Clinical Hospital of the Moscow City Health Department State-Financed (Unknown)
Responsible Party: Sponsor-Investigator, Anna Vlasova, PhD, chief of Clinical Pharmacology department, National Medical Research Center for Children's Health, Russian Federation
Organization: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Other Study IDs: 07819001
Record Dates: First submitted 2019-10-09; First posted 2019-10-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Drug Therapy
Keywords: neonates; antimicrobial pharmacotherapy; pharmacotherapy adverse events; neonatal Intensive Care Unit; safety
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genotyping will be performed using the modification option of VeriDose® Core Panel (VeriDose and Agena Bioscience are registered trademarks of Agena Bioscience, Inc.).
  VeriDose® Core Panel provides the detection of the most relevant variants in the key genes involved in drug metabolism pathways: Pg-s gene ABCB1, APOE, CYP1A2, CYP2B6, CYP2C19, CYP2D6, CYP3A4, CYP3A5, DRD2, F2, F5, GLP1R, MTHFR, OPRM1, PNPLA5, SLCO1B1, SULT4A1, VKORC1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1 (0-17 years): We will observe the treatment course in ICU pediatric patients, register adverse events (AEs) and serious adverse events (SAEs) if occur, and assess patient health status at the end of the performed therapy.
  Interventions: Other: Pharmacogenetic test

INTERVENTIONS:
Other: Pharmacogenetic test — Buccal swabs are a relatively non-invasive way to collect deoxyribonucleic acid (DNA) samples for testing. A buccal swab will be performed to collect DNA from the cells on the inside of a subject's cheek for phenotyping of CYP3A4.
  Other Names: Buccal swabs for pharmacogenetic testing; buccal smear

SUMMARY:
Changes in the metabolic ability of cytochrome P-450 during child development can affect both bioavailability and elimination depending on the involvement of intestinal and hepatic metabolic processes. The age-related variability of cytochrome P-450 isoenzymes in children has been described since 2010. The variability in the development of the activity of specific cytochrome P-450 isoenzymes illustrates why the pharmacogenetic features of the medicine use at different age periods should be studied for individual drugs. This will provide an understanding of the mechanisms for preventing adverse events appearing in pediatric intensive care units while more common antimicrobial pharmacotherapy is administered. Improved knowledge of the pharmacogenetic characteristics of cytochrome P-450 and the unintended consequences of modulation of its isoenzymes could provide an understanding of the susceptibility to adverse events in children in critical conditions staying at Intensive Care unit (ICU).

DETAILED DESCRIPTION:
An observational prospective multidirectional study on the safety of antimicrobial pharmacotherapy in ICU children aged 0-17. The endpoints of the safety assessment are the frequency of adverse events with antimicrobial agents (AMA); electrocardiography (ECG), fibrinogen concentration, international normalized ratio (INR) and prothrombin index (IPT) at screening and at the end of the treatment course, and pharmacogenetic indicators (a more detailed study of the safety profile). A demonstration of the effectiveness of each of these comparisons of inequality will be based on the hypothesis testing approach, according to which the null hypothesis concludes that there is no difference between groups receiving different AMA combinations for the endpoint of interest; and an alternative hypothesis supposes a difference between treatment groups receiving different AMA combinations. Changes in the sequential organ failure assessment (SOFA) scale in dynamics compared to the baseline will be analyzed using the Mixed-Effect Model Repeated Measure (MMRM) model which assume the baseline, gender, age, AMA combination, and the duration of the AMA course. For a population of subjects aged 0-3 months, the analysis will be performed using the analysis of covariance (ANCOVA) model with the effects of INR, fibrinogen, and IPT values at the initial level for gender, age, and AMA combination in the treatment groups.

To assess the secondary endpoint for the general population - the frequency and timing of the transition to de-escalation at ICU, cluster analysis will be conducted to identify the relationship of specific AMA combinations with the possibility of de-escalation in ICU children.

Studies will be conducted to reveal the relationship in gene polymorphism encoding isoenzymes of the cytochrome P-450 biotransformation, and the relationship between the activity of transport proteins with the indicators of effectiveness and safety of antimicrobial pharmacotherapy. The lack of pharmacological safety studies in children administered medicine combinations to overcome pan-resistant gram-negative infection provides relevant prerequisites for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Intensive Care Unit (ICU) patient;
2. Community-acquired infections with risk factors for multidrug-resistant pathogens (risk factors for extended-spectrum β-lactamase (ESBL) - type II;
3. Nosocomial infections - type III:

   * IIIa: hospitalized during the period of 90 days, without prior antimicrobial agent (AMA) therapy outside the ICU (risk factors for ESBL);
   * IIIb: prolonged hospitalization (> 7 days) and/or stay at ICU for more than 3 days and/or previous AMA therapy (risk factors for ESBL, carbenicillin-resistant (CARB-R), nonfermenting Gram-negative bacteria (NFGNB), methicillin-resistant Staphylococcus aureus (MRSA));
4. Nosocomial infections with a risk of invasive candidiasis - type IV (candida score ≥2 points);
5. Written informed consent for medical intervention signed by at least one parent or caregiver (legal guardian) or informed consent of a patient under 15 years of age;
6. Written informed consent for pharmacogenetic research signed by at least one parent or caregiver (legal guardian) or informed consent of a patient under 15 years of age.

Exclusion Criteria:

1. Type I: patients with community-acquired infections and without risk factors for multidrug-resistant pathogens, without hospitalization during the previous 90 days;
2. Previous/concomitant therapy is not significant;
3. Children in the ward: children under guardianship are not eligible.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll the participants from the patients of the Intensive Care Unit at Morozov Children's City Clinical Hospital of the Moscow City Health Department, Moscow, Russian Federation.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Adverse events frequency | From baseline until the date of first documented progression, assessed up to 1 month
  Registered adverse events in participants during the treatment course
ECG QT Interval change | Change from screening QT Interval at 1 month
  Assessment of QT Interval change at the end of the AMA course comparing with screening measurement

CONTACTS AND LOCATIONS:
Overall Officials: Anna Vlasova, PhD, MD, Principal Investigator — Morozov Children's City Clinical Hospital of the Moscow City Health Department
Locations (1):
- Morozov Children's City Clinical Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available partially upon a request.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data Access Requests will be reviewed by the Independent Local Review Board. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Ward RM, Benjamin D, Barrett JS, Allegaert K, Portman R, Davis JM, Turner MA. Safety, dosing, and pharmaceutical quality for studies that evaluate medicinal products (including biological products) in neonates. Pediatr Res. 2017 May;81(5):692-711. doi: 10.1038/pr.2016.221. Epub 2016 Nov 3. PMID 28248319
- [Result] Martinez Tadeo JA, Perez Rodriguez E, Almeida Sanchez Z, Callero Viera A, Garcia Robaina JC. No Cross-Reactivity With Cephalosporins in Patients With Penicillin Allergy. J Investig Allergol Clin Immunol. 2015;25(3):216-7. No abstract available. PMID 26182689
- [Result] Ball P. Quinolone-induced QT interval prolongation: a not-so-unexpected class effect. J Antimicrob Chemother. 2000 May;45(5):557-9. doi: 10.1093/jac/45.5.557. No abstract available. PMID 10797074
- [Result] Schliamser SE, Broholm KA, Liljedahl AL, Norrby SR. Comparative neurotoxicity of benzylpenicillin, imipenem/cilastatin and FCE 22101, a new injectible penem. J Antimicrob Chemother. 1988 Nov;22(5):687-95. doi: 10.1093/jac/22.5.687. PMID 3209527
- [Result] Odio CM, Puig JR, Feris JM, Khan WN, Rodriguez WJ, McCracken GH Jr, Bradley JS. Prospective, randomized, investigator-blinded study of the efficacy and safety of meropenem vs. cefotaxime therapy in bacterial meningitis in children. Meropenem Meningitis Study Group. Pediatr Infect Dis J. 1999 Jul;18(7):581-90. doi: 10.1097/00006454-199907000-00004. PMID 10440432
- [Result] Cui L, Kasegawa H, Murakami Y, Hanaki H, Hiramatsu K. Postoperative toxic shock syndrome caused by a highly virulent methicillin-resistant Staphylococcus aureus strain. Scand J Infect Dis. 1999;31(2):208-9. doi: 10.1080/003655499750006326. PMID 10447337
- [Result] Norrby SR. Carbapenems in serious infections: a risk-benefit assessment. Drug Saf. 2000 Mar;22(3):191-4. doi: 10.2165/00002018-200022030-00003. PMID 10738843
- [Result] Winston DJ, Lazarus HM, Beveridge RA, Hathorn JW, Gucalp R, Ramphal R, Chow AW, Ho WG, Horn R, Feld R, Louie TJ, Territo MC, Blumer JL, Tack KJ. Randomized, double-blind, multicenter trial comparing clinafloxacin with imipenem as empirical monotherapy for febrile granulocytopenic patients. Clin Infect Dis. 2001 Feb 1;32(3):381-90. doi: 10.1086/318500. Epub 2001 Jan 30. PMID 11170945
- [Result] Karadeniz C, Oguz A, Canter B, Serdaroglu A. Incidence of seizures in pediatric cancer patients treated with imipenem/cilastatin. Pediatr Hematol Oncol. 2000 Oct-Nov;17(7):585-90. doi: 10.1080/08880010050122852. PMID 11033734
- [Result] Smith RG. Penicillin and cephalosporin drug allergies: a paradigm shift. J Am Podiatr Med Assoc. 2008 Nov-Dec;98(6):479-88. doi: 10.7547/0980479. PMID 19017859
- [Result] Laughon MM, Avant D, Tripathi N, Hornik CP, Cohen-Wolkowiez M, Clark RH, Smith PB, Rodriguez W. Drug labeling and exposure in neonates. JAMA Pediatr. 2014 Feb;168(2):130-6. doi: 10.1001/jamapediatrics.2013.4208. PMID 24322269
- [Result] Setiawan E, Suwannoi L, Montakantikul P, Chindavijak B. Optimization of Intermittent Vancomycin Dosage Regimens for Thai Critically Ill Population Infected by MRSA in the Era of the "MIC Creep" Phenomenon. Acta Med Indones. 2019 Jan;51(1):10-18. PMID 31073101
- [Result] Leon C, Ruiz-Santana S, Saavedra P, Almirante B, Nolla-Salas J, Alvarez-Lerma F, Garnacho-Montero J, Leon MA; EPCAN Study Group. A bedside scoring system ("Candida score") for early antifungal treatment in nonneutropenic critically ill patients with Candida colonization. Crit Care Med. 2006 Mar;34(3):730-7. doi: 10.1097/01.CCM.0000202208.37364.7D. PMID 16505659
- [Result] Prot-Labarthe S, Weil T, Angoulvant F, Boulkedid R, Alberti C, Bourdon O. POPI (Pediatrics: Omission of Prescriptions and Inappropriate prescriptions): development of a tool to identify inappropriate prescribing. PLoS One. 2014 Jun 30;9(6):e101171. doi: 10.1371/journal.pone.0101171. eCollection 2014. PMID 24978045
- [Result] Yahav D, Lador A, Paul M, Leibovici L. Efficacy and safety of tigecycline: a systematic review and meta-analysis. J Antimicrob Chemother. 2011 Sep;66(9):1963-71. doi: 10.1093/jac/dkr242. Epub 2011 Jun 18. PMID 21685488
- [Result] McGovern PC, Wible M, El-Tahtawy A, Biswas P, Meyer RD. All-cause mortality imbalance in the tigecycline phase 3 and 4 clinical trials. Int J Antimicrob Agents. 2013 May;41(5):463-7. doi: 10.1016/j.ijantimicag.2013.01.020. Epub 2013 Mar 26. PMID 23537581
- [Result] Ellis-Grosse EJ, Babinchak T, Dartois N, Rose G, Loh E; Tigecycline 300 cSSSI Study Group; Tigecycline 305 cSSSI Study Group. The efficacy and safety of tigecycline in the treatment of skin and skin-structure infections: results of 2 double-blind phase 3 comparison studies with vancomycin-aztreonam. Clin Infect Dis. 2005 Sep 1;41 Suppl 5:S341-53. doi: 10.1086/431675. PMID 16080072
- [Result] Baietto L, Corcione S, Pacini G, Perri GD, D'Avolio A, De Rosa FG. A 30-years review on pharmacokinetics of antibiotics: is the right time for pharmacogenetics? Curr Drug Metab. 2014;15(6):581-98. doi: 10.2174/1389200215666140605130935. PMID 24909419
- [Result] Kim K, Johnson JA, Derendorf H. Differences in drug pharmacokinetics between East Asians and Caucasians and the role of genetic polymorphisms. J Clin Pharmacol. 2004 Oct;44(10):1083-105. doi: 10.1177/0091270004268128. PMID 15342610
- [Result] Matthews HW. Racial, ethnic and gender differences in response to medicines. Drug Metabol Drug Interact. 1995;12(2):77-91. doi: 10.1515/dmdi.1995.12.2.77. PMID 8591695
- See also: Karaiskos I, Barmpouti E, Ioannidis K, et al. Hypofibrinogenaemia associated with the administration of tigecycline. Conference Paper (poster). Conference: 24th ECCMID; 2014, Barcelona, Spain. doi: 10.13140/2.1.2337.2163. — https://www.researchgate.net/publication/265553167_Hypofibrinogenaemia_associated_with_the_administration_of_tigecycline